CLINICAL TRIAL: NCT05994456
Title: Neoadjuvant Toripalimab in the Treatment of Locally Advanced dMMR/MSI-H Gastric or Gastroesophageal Junction Adenocarcinoma：an Open-label, Single-arm，Multi-center，Phase II Trial
Brief Title: Neoadjuvant Toripalimab for dMMR/MSI-H Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dong sheng Zhang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP001
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Gastric or Gastroesophageal Junction Adenocarcinoma
Keywords: dMMR/MSI-H; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Immune Checkpoint Inhibitors; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 inhibitor (Experimental): Neoadjuvant therapy with PD-1 inhibitor (Toripalimab)
  Interventions: Drug: PD-1 inhibitor

INTERVENTIONS:
Drug: PD-1 inhibitor — 240mg, Q3W. The opportunity for surgery was evaluated after 2 cycles of treatment and surgical treatment was performed after 2-4 cycles of treatment. Postoperatively, adjuvant therapy was continued according to the neoadjuvant regimen, and direct treatment met the criteria for termination of treatment.
  Other Names: Toripalimab

SUMMARY:
This is a single-center, open phase II clinical trial to evaluate the tolerability, safety and efficacy of toriparib monotherapy in the treatment of locally advanced dMMR/MSI-H gastric or gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
In this phase II study, eligible patients are enrolled to receive toripalimab 240mg, ivdrip, Q3W to evaluate the anti-tumor efficacy and safety. After 2 and 4 cycles of toripalimab treatment, tumors are assessed, and patients are assigned to receive surgery or withdraw from study according to their anti-tumor efficacy. For patients withdrawing from study, routine treatment would be given. For patients staying in study, toripalimab would be administered for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, regardless of gender 2. Patients with histologically or cytologically confirmed adenocarcinoma of the stomach or gastroesophageal junction and confirmed dMMR or MSI-H 3. Preoperative CT or MRI staging meeting the following criteria: T2 and above, with or without lymph node involvement, without clear distant metastasis 4. ECOG score of 0-1. 5. Expected survival ≥ 2 years. 6. Good organ function (no blood transfusion, no hematopoietic stimulating factor, no albumin or blood product transfusion within 14 days prior to the examination).

1. Platelet (PLT) count ≥ 90*109/L.
2. Neutrophil count (ANC) ≥ 1.5*109/L.
3. Hemoglobin (Hb) level ≥ 9.0 g/dl.
4. International normalized ratio (INR) ≤ 1.5.
5. Prothrombin time (PT) and active partial thromboplastin time (APTT) ≤ 1.5 x ULN.
6. Glycated hemoglobin (HbA1c) <7.5%.
7. Total bilirubin (TBIL) level ≤ 1.5 times the upper limit of normal (ULN).
8. Alanine amino transaminase (ALT) and aspartate amino transaminase (AST) levels ≤ 2.5 x ULN.
9. Serum creatinine (Cr) level ≤ 1.5 x ULN and creatinine clearance ≥ 60 ml/min.
10. Thyrotropin (TSH) ≤ ULN; serum free thyroid hormone (T4) normal; serum free triiodothyronine (T3) normal; (except for those who have received previous thyroid surgery or have a history of head and neck radiotherapy)
11. Serum amylase ≤ 1.5 x ULN.
12. Lipase ≤ 1.5×ULN. 7. Women of childbearing age must have a negative pregnancy test and must use contraception and avoid breastfeeding during the study and for 3 months after the last dose; male subjects must agree to use contraception during the study and for 3 months after the last dose.

8.Be able to understand and willing to sign a written informed consent form.

Exclusion Criteria:

1. Previously received chemotherapy, radiotherapy or immunotherapy for gastric cancer
2. Previously diagnosed any other malignancy with a primary site or histological type different from gastric cancer within 5 years prior to study entry, except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
3. With known hypersensitivity to the study drug or excipients, or to similar drugs
4. Received major surgery or open biopsy, or had a major trauma within 4 weeks prior to the start of study treatment
5. Received immunosuppressive drugs (excluding inhaled corticosteroids or ≤10 mg/day prednisone or equivalent pharmacophysiologic doses of other systemic steroids) within 2 weeks prior to the start of study treatment
6. Planned live attenuated vaccination within 4 weeks prior to the start of study treatment or during the study period
7. Inability to discontinue CYP3A4 inducers or inhibitors within 1 week prior to the start of study treatment and during the study period
8. Presence of any autoimmune disease or history of autoimmune disease.
9. Human immunodeficiency virus (HIV) infection (HIV antibody positive), or active hepatitis C virus (HCV) infection (HCV antibody positive), or active hepatitis B virus (HBV) infection (HBsAg positive and HBV-DNA ≥ 2000 IU/ml copies/ml)), or other serious infection requiring antibiotics for systemic therapy, or during screening/study Unexplained temperature >38.5°C prior to the start of treatment.
10. Presence of the following diseases within 6 months prior to the start of study treatment: myocardial infarction, severe/unstable angina, NYHA class 2 or higher congestive heart failure, poorly controlled arrhythmias, etc.
11. Non-well-controlled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg under optimal treatment)
12. Arterial/venous thrombotic events such as cerebrovascular accidents (transient ischemic attack, cerebral hemorrhage, cerebral infarction, etc.), deep vein thrombosis, vasculitis, etc. within 3 months prior to the start of study treatment
13. Urine routine suggesting urine protein up to +++ and confirmed 24-hour urine protein quantification up to 1.0g.
14. The presence of a history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
15. Seizures requiring medication (e.g., steroids or antiepileptic drugs) for treatment.
16. Presence of a history of substance abuse, drug use, or alcohol dependence. Patients with other serious, acute or chronic medical conditions that may increase the risk of study participation and study medication, or that may interfere with the interpretation of study results, and who are judged by the investigator to be unsuitable for participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission (pCR) rates | 12 weeks
  Percentage of patients who achieve pathological complete remission (pCR)

SECONDARY OUTCOMES:
R0 resection rates | 12 weeks
  The proportion of patients experiencing a R0 resection
three-year disease-free survival rate, DFS | 3 years
  Percentage of patients who achieve disease-free survival lasting for more than three years
three-year Overall survival rate,OS | 3 years
  Percentage of patients who achieve survival for more than two years
Incidence of Treatment-Related Adverse Events | 3 years
  Number of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Zhang, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China